CLINICAL TRIAL: NCT02035475
Title: A Pilot Clinical Trial for the Prevention of Lymphoceles After Robotic Pelvic Lymph Node Dissections for Prostate Malignancies Using the da Vinci® EndoWrist® One™ Vessel Sealer
Brief Title: Prevention of Lymphoceles After Robotic PLND
Acronym: PLND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OhioHealth (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Principal Investigator, Ronney Abaza, Medical Director Robotic Surgery, OhioHealth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: OH1-13-00471
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-04

CONDITIONS: Lymphoceles; Prostate Cancer
Keywords: Prevention; Pelvic Lymph Node Dissection; Lymphoceles; Prostate Malignancies; daVinci; Vessel Sealer; EndoWrist One
MeSH Terms: conditions — Lymphocele; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intuitive Vessel Sealer (Active Comparator): Investigators intend to use this device unilaterally so the contralateral side can serve as an internal control.
  Interventions: Device: Intuitive Vessel Sealer
- Maryland Bipolar Cautery (Active Comparator): Investigators intend to use this device unilaterally so the contralateral side can serve as an internal control.
  Interventions: Device: Intuitive Vessel Sealer

INTERVENTIONS:
Device: Intuitive Vessel Sealer — Investigators intend to use this device unilaterally so the contralateral side can serve as an internal control.
  Other Names: EndoWrist One Vessel Sealer

SUMMARY:
The EndoWrist One Vessel Sealer is a bipolar electrosurgical instrument for use with the da Vinci Si robotic surgical system. It is intended for bipolar coagulation and mechanical transection of vessels up to 7 mm in diameter and tissue bundles that fit within the jaws of the instrument. Their use in this study will be to perform tissue transection during PLND such that the intended use is within the FDA-approved domain for this instrument. Investigators intend to identify whether its use for PLND reduces lymphoceles given that the device is known to seal vessels up to 7 mm, which is much larger than lymphatic vessels encountered during PLND. Because the instrument is new and has been FDA approved for less than one year, there is no published literature regarding its use to date.

Our hypothesis is that using the Vessel Sealer on a single side of the pelvis will reduce the incidence of screening detected lymphoceles on that side. Investigators propose a total sample size of 120 patients.

DETAILED DESCRIPTION:
Investigators propose a prospective, randomized, single-blinded study of patients diagnosed with pelvic cancer who are electing to undergo robotic surgery with PLND. The patients in our trial will be pelvic cancer patients at risk for lymphocele after PLND. Given the safe nature of the product and the patient's risk for lymphocele after PLND and subsequent potential morbidity, there is justification to give patients the option for inclusion in the study. Investigators intend to determine whether the rate of lymphocele formation after PLND at the time of robotic pelvic cancer surgery can be reduced by using the robotic Vessel Sealer unilaterally for the lymph node dissection. The side of the pelvis of each patient will be randomly selected by Excel's® random number function "RAND()" to receive the Vessel Sealer dissection. Investigators intend to use this device unilaterally so the contralateral side can serve as an internal control and eliminate patient specific confounding variables such as BMI, and surgeon specific factors such as degree and method of hemostasis utilized by each surgeon. In addition, Dr. Abaza will be the only surgeon performing these procedures, eliminating variation in technique between surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Candidate scheduled to undergo robotic prostatectomy surgery with PLND

Exclusion Criteria:

* Age < 18
* Unable to give informed consent
* Non-English speaking
* Not a candidate for robotic surgery for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronney Abaza, MD, FACS, Principal Investigator — OhioHealth
Locations (1):
- Dublin Methodist Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Abaza R, Henderson SJ, Martinez O. Robotic Vessel Sealer Device for Lymphocele Prevention After Pelvic Lymphadenectomy: Results of a Randomized Trial. J Laparoendosc Adv Surg Tech A. 2022 Jul;32(7):721-726. doi: 10.1089/lap.2021.0531. Epub 2021 Oct 22. PMID 34677080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prostatectomy patients were recruited from a single robotic urologists office, between 1/15/13 and 5/12/14. The final followup visit was completed on 12/18/14.
Pre-assignment Details: Participants must be eligible for robotic procedures.
Period: Overall Study
Arm/Group | Intuitive Vessel Sealer
Started | 120 (120 subjects were consented for participation in the study.)
Completed | 114 (Six subjects did not complete the study due to withdrawal of consent.)
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Equipment Error | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intuitive Vessel Sealer
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 114

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Lymphoceles
Description: Identify whether the use of the Vessel Sealer for PLND reduces the incidence of screening detected lymphoceles via CT scan of the pelvis by comparing the Vessel Sealer side of the pelvis with the control side of the pelvis.
Time Frame: 4 months
Population: Lymphoceles were identified by CT scan at 3 months post surgery.
Measure: Number; unit: participants
Groups:
- EndoWrist 1 Vessel Sealer: Investigators intend to use this device unilaterally so the contralateral side can serve as an internal control.
  The EndoWrist 1 Vessel Sealer was utilized on one side of the body, with each participant receiving both treatments, one each side.
- Fenestrated Maryland BiPolar Instrument: The Fenestrated Maryland BiPolar Instrument was utilized on one side of the body, with each participant receiving both treatments, one each side.
Arm/Group | EndoWrist 1 Vessel Sealer | Fenestrated Maryland BiPolar Instrument
Number analyzed (Participants) | 114 | 114
participants
  Lymphoceles | 10 | 12
  No Lymphoceles | 104 | 102
Statistical Analysis 1: Comparison: EndoWrist 1 Vessel Sealer vs Fenestrated Maryland BiPolar Instrument; The null hypothesis is that there is no difference in the incidence of detected lymphoceles whether the EndoWrist 1 Vessel Sealer or the Fenestrated Maryland BiPolar Instrument were used; Test type: Superiority or Other; p = 0.412, McNemar

2. Secondary Outcome: Surgical Complications
Description: Evaluate perioperative and postoperative surgical outcomes at 4 months after surgery. Possible outcomes include "no complications" (0), "minor complications" (1), and "major complications" (2).
Time Frame: 4 months
Measure: Number; unit: participants
Groups:
- Study Participants: Investigators intend to use this device unilaterally so the contralateral side can serve as an internal control.
  Intuitive Vessel Sealer: Investigators intend to use this device unilaterally so the contralateral side can serve as an internal control.
Arm/Group | Study Participants
Number analyzed (Participants) | 114
participants | 3

ADVERSE EVENTS:
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 3/114
Other Adverse Events (participants affected / at risk) | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=114)
Rehospitalization (General disorders) | 1 (1) — Rehospitalization due to fever and back pain.
Bilateral Pulmonary Embolisms (Blood and lymphatic system disorders) | 1 (1) — Shortness of breath. ER visit-CT angioplasty with thrombolysis and IVC filter placement with extended hospital (2 day) stay.
Prolonged existing hospitalization (General disorders) | 2 (2) — Post-operative course complicated by syncope (likely vasovagal in context of pain), SOB, Ileus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No